CLINICAL TRIAL: NCT05423145
Title: Self-Administered Acupressure for Veterans With Chronic Back Pain: A Multisite Evaluation of Effectiveness and Implementation
Brief Title: Self-Administered Acupressure for Veterans With Chronic Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 20-242; 1I01HX003302-01A2 (NIH)
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: acupressure; complementary therapies
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: two groups, intervention and wait list control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and analyst conducting the main analysis will be masked. The participants and project staff will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupressure intervention (Experimental): Receives access to the acupressure intervention
  Interventions: Behavioral: self-administered acupressure
- wait list control (No Intervention): No access to the acupressure intervention during the study period

INTERVENTIONS:
Behavioral: self-administered acupressure — The acupressure intervention is self-administered. The intervention group receives an app that instructs them on how to perform a stimulating acupressure protocol, consisting of six acupoints with four of the acupoints performed on both the left and the right sides of the body for a total of ten points. Each of the ten acupoints is to be stimulated for 3 minutes per point for a total treatment time of 30 minutes daily for 6 weeks.
  Arms: acupressure intervention

SUMMARY:
Many Veterans experience chronic pain, with back pain the most commonly reported condition. The Veterans Health Administration (VHA) is moving from reliance on medications to an approach in which non-medication interventions, including complementary and integrative health treatments, are now a first line of care. Acupressure, a Traditional Chinese Medicine technique derived from acupuncture, is emerging as a potentially effective approach for treating several chronic pain conditions and could prove beneficial in helping Veterans manage their chronic low back pain.

This study will determine the effectiveness of self-administered acupressure to treat chronic low back pain. 300 Veterans will be invited to participate in the study. All participants will be asked to attend an introduction to acupressure class and complete a survey when they join the study and again at 6 weeks and 10 weeks. The survey measures assess important outcomes, such as how pain interferes with daily function, as well as other areas that can be affected by pain such as fatigue and sleep quality. After completing the first survey, half of the participants will receive a tablet computer with an app that shows them how to self-administer acupressure for low back pain and will be asked to do daily acupressure sessions for the next 6 weeks. The other half of the participants will receive the tablet computer with the app approximately 10 weeks after completing the final survey based assessment. The investigators anticipate that outcomes will be improved after 6 weeks of acupressure practice, and these improvements will persist for the following 4 weeks.

DETAILED DESCRIPTION:
This is a hybrid Type 1 effectiveness implementation study. The primary aim is to conduct a 2-group, randomized controlled trial to examine the effectiveness of stimulating acupressure compared to a waitlist control group for Veterans with chronic low back pain. Study participants will include Veterans Health Administration patients within the VA Ann Arbor Healthcare System who suffer from chronic low back pain and are interested in trying acupressure as a form of pain management. The second aim is to assess facilitators and barriers to implementing this type of acupressure program in VHA.

Specifically, this study will determine the effectiveness of a 6-week self-administered acupressure protocol on outcomes of pain interference, fatigue, sleep quality, and disability, at 6- and 10-weeks post baseline compared to a waitlist control group. The investigators hypothesize that outcomes will be improved from baseline for Veterans after 6 weeks of acupressure practice, and improvements will persist for the following 4 weeks. Intervention effects will be moderated by opioid use at baseline, age, sex, and baseline pain interference.

The study will recruit and enroll 300 Veterans with chronic low back pain, who will be randomized into one of two study arms: stimulating acupressure or a waitlist control group. These Veterans will be recruited in multiple ways, including through Whole Health classes offered at the study facilities, provider referral and proactive outreach, with potentially eligible participants identified using electronic health record data available through the VHA's Corporate Data Warehouse. All participants will attend an introductory acupressure class, conducted either virtually or in person, that provides a general overview of acupressure for chronic back pain, demonstrates how to find an acupressure point and how much pressure to apply.

After completing the consent process and a baseline survey, participants will be randomized to the acupressure intervention or waitlist control group. Participants will be allocated into groups in a 1:1 ratio by block randomization with mixed block sizes and stratified by sex to ensure balance of females and males across groups. Participants randomized to the intervention will then receive a tablet computer with an app that provides specific instructions on how to self-administer stimulating acupressure and identify acupressure points for treating back pain. Intervention participants will be asked to follow a 6-week protocol that involves performing acupressure once per day, for approximately 30 minutes, guided by the app. After 6 weeks, they will be asked to stop acupressure for 4 weeks so persisting effects can be determined. Participants in the waitlist control group will receive a tablet with the app at the end of 10 weeks. Survey based outcome assessments will be conducted at 6 weeks and 10 weeks.

The ultimate goal of this study is to identify effective and accessible non-pharmacological treatments for chronic pain, which are critically needed both inside and outside VHA.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled at VA Ann Arbor Healthcare System
* non-specific low back pain confirmed through electronic medical records (i.e., ICD-10 codes: M54.5, M54.40, 41, 42, M54.89)
* reported pain severity of 4/10 that has persisted for at least 3 months and present on most days
* medically stable (no hospitalizations in the past month lasting 3 or more days)
* no changes in pain medication regimen in past 4 weeks
* no planned surgery or injections for back pain during the next 10 weeks

Exclusion Criteria:

* pregnant
* had back surgery in the past 2 years
* received acupuncture or acupressure in past 3 months
* evidence of cognitive impairment that could interfere with the ability to provide consent and follow the study protocol (defined as a score of 3 using the Callahan et al. 6-item screener)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
change in PROMIS 6b pain interference scale | baseline to 6 weeks (end of active treatment) and 10 weeks (sustainability)
  The Pain Interference Scale provides an assessment of the impact of pain on several aspects of functioning, including social and emotional processes as well as physical function (e.g., how much did pain interfere with your day to day activities) based on 6 items rated on a scale of 1 (not at all) to 5 (very much). Final scores are given as T-scores, with higher scores representing greater interference (worse function). PROMIS scores are a t-score representing relationships with an estimated population average collected on a general US sample of adults as well as clinical samples. On this t distribution, 50 represents the population average with a standard deviation of 10. Thus, a score of 60 represents a score that is 1 standard deviation above the US national average, and a 40 represents a score that is 1 standard deviation below the national average.

SECONDARY OUTCOMES:
change in PROMIS 8a fatigue scale | baseline to 6 weeks (end of active treatment) and 10 weeks (sustainability)
  The fatigue scale consists of 8 items that assess the degree and impact of fatigue with each item rated on a scale of 1 (not at all) to 5 (very much). Final scores are given as T-scores, with higher scores representing worse fatigue. PROMIS scores are a t-score representing relationships with an estimated population average collected on a general US sample of adults as well as clinical samples. On this t distribution, 50 represents the population average with a standard deviation of 10. Thus, a score of 60 represents a score that is 1 standard deviation above the US national average, and a 40 represents a score that is 1 standard deviation below the national average.
change in PROMIS 8b sleep disturbance scale | baseline to 6 weeks (end of active treatment) and 10 weeks (sustainability)
  The sleep disturbance scale consists of 8 items that assess sleep quality with each item rated on a scale of 1 (not at all) to 5 (very much). Final scores are given as T-scores, with higher scores representing worse sleep disturbance. PROMIS scores are a t-score representing relationships with an estimated population average collected on a general US sample of adults as well as clinical samples. On this t distribution, 50 represents the population average with a standard deviation of 10. Thus, a score of 60 represents a score that is 1 standard deviation above the US national average, and a 40 represents a score that is 1 standard deviation below the national average.
change in Roland Morris Disability scale | baseline to 6 weeks (end of active treatment) and 10 weeks (sustainability)
  The Roland Morris disability scale is an assement of back pain specific disability based on the total number of items checked, ranging from a minimum of 0 to a maximum of 24, with higher scores indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Krein, PhD RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy SL, Zick SM, Harris RE, Smith SN, Sen A, Alexander NB, Caldararo J, Roman P, Firsht E, Belancourt P, Maciasz R, Perzhinsky J, Mitchinson A, Krein SL. Self-administered acupressure for veterans with chronic back pain: Study design and methodology of a type 1 hybrid effectiveness implementation randomized controlled trial. Contemp Clin Trials. 2023 Jul;130:107232. doi: 10.1016/j.cct.2023.107232. Epub 2023 May 18. PMID 37207810

DOCUMENTS (1):
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05423145/ICF_000.pdf